CLINICAL TRIAL: NCT06350526
Title: Radiological Characterization of Pulmonary Involvement in Patients With Hematological Diseases
Status: Completed | Type: Observational
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Asmaa Nady Hussein, Lecturer of Internal Medicine, New Valley University
Other Study IDs: PULMHEMA
Record Dates: First submitted 2024-02-01; First posted 2024-04-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Blood Cell Count; Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patient admitted with hematological disease and pulmonary manifestations
  Interventions: Diagnostic Test: Complete Blood Count; Diagnostic Test: C-reactive protein; Diagnostic Test: O2 saturation; Diagnostic Test: Serum ferritin and D-dimer; Diagnostic Test: Liver and renal function tests; Diagnostic Test: Lactate dehydrogenase; Diagnostic Test: coronavirus (SARS-CoV-2) swab; Radiation: CT chest

INTERVENTIONS:
Diagnostic Test: Complete Blood Count — blood sample
Diagnostic Test: C-reactive protein — serum sample
Diagnostic Test: O2 saturation — blood sample
Diagnostic Test: Serum ferritin and D-dimer — Blood sample
Diagnostic Test: Liver and renal function tests — Blood sample
Diagnostic Test: Lactate dehydrogenase — Blood sample
Diagnostic Test: coronavirus (SARS-CoV-2) swab — Throat swab
Radiation: CT chest — Radiation

SUMMARY:
Hematologic malignancies are heterogeneous groups of neoplasia, with frequent pulmonary complications. These complications may be secondary to the patient's comorbidities, to the hemopathy itself, or its treatments. Divided into infectious and non-infectious complications, the etiologies are numerous and varied. This makes the diagnostic approach complex for the clinicians

DETAILED DESCRIPTION:
Although infectious processes of the lungs are common in these immunosuppressed patient collectives, non-infectious causes account for up to half of the pulmonary manifestations found in hematologic malignancies. Besides the frequent infections including opportunistic pathogens, a broad differential diagnosis including drug-induced lung injury by cytostatic substances, cytokines, and innovative immunotherapeutic agents, rarer transfusion of blood products, and intrathoracic manifestations of the hematologic malignancy itself, must be kept in mind. Finally, vascular complications can also lead to pulmonary reactions. Early and consistent diagnostics and treatment of bronchopulmonary, intrathoracic, and vascular complications within the framework of hematologic systemic diseases can be essential for the patient's prognosis. Up to 25% of patients with profound neutropenia lasting for >10 days develop lung infiltrates, which frequently do not respond to broad-spectrum antibacterial therapy. While a causative pathogen remains undetected in most cases, Aspergillus spp., Pneumocystis jirovecii, multi-resistant Gram-negative pathogens, mycobacteria or respiratory viruses may be involved. In at-risk patients who have received trimethoprim-sulfamethoxazole (TMP/SMX) prophylaxis, filamentous fungal pathogens appear to be predominant, yet commonly not proven at the time of treatment initiation.

In patients who do not improve rapidly with first-line therapy with broad spectrum antibiotics, cross-sectional thoracic CT imaging is essential. It provides much better definition of the pattern of radiological changes that includes three main groups: consolidation, nodules (micro- and macro-), and diffuse changes, as ground glass pattern. Discuss these radiological patterns and how this guides the appropriate initial investigations and treatment options will be of a great value to be followed.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years or older diagnosed with hematological diseases and documented pulmonary manifestations during their disease course

Exclusion Criteria:

1. Patients aged under 18 years.
2. Patients without demonstrable evidence of lung involvement.
3. Patients with incomplete medical records or insufficient data to analyze.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older diagnosed with hematological diseases and documented pulmonary manifestations during their disease course will be included in this retrospective study. Data from their medical records will be analyzed by a team of hematologists, pulmonologists, and radiologists.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Number of patients who had certain radiological patterns associated with pulmonary complications in patients diagnosed with various hematological diseases | Once through the study

SECONDARY OUTCOMES:
Number of patients who developed complications | Once through the study

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Messe R, Soccal PM, Bergeron A. [Diagnostic approach to pulmonary complications in patients with hematologic malignancy]. Rev Med Suisse. 2021 Nov 17;17(759):1984-1990. French. PMID 34787973
- [Background] Stecher SS, Lippl S, Stemmler HJ, Schreiber J. [Lung involvement in hematologic systemic diseases]. Internist (Berl). 2018 Sep;59(9):886-897. doi: 10.1007/s00108-018-0471-9. German. PMID 30046891
- [Background] Maschmeyer G, Carratala J, Buchheidt D, Hamprecht A, Heussel CP, Kahl C, Lorenz J, Neumann S, Rieger C, Ruhnke M, Salwender H, Schmidt-Hieber M, Azoulay E. Diagnosis and antimicrobial therapy of lung infiltrates in febrile neutropenic patients (allogeneic SCT excluded): updated guidelines of the Infectious Diseases Working Party (AGIHO) of the German Society of Hematology and Medical Oncology (DGHO). Ann Oncol. 2015 Jan;26(1):21-33. doi: 10.1093/annonc/mdu192. Epub 2014 May 15. PMID 24833776
- [Background] Periselneris J, Brown JS. A clinical approach to respiratory disease in patients with hematological malignancy, with a focus on respiratory infection. Med Mycol. 2019 Jun 1;57(Supplement_3):S318-S327. doi: 10.1093/mmy/myy138. PMID 31292655